CLINICAL TRIAL: NCT06383286
Title: The Relationship Between Physical Activity Levels and Anxiety, Depression, Stress of Disabled Athletes Who Prepared for Paralympic Games
Brief Title: The Relationship Between Physical Activity Levels and Anxiety, Depression, Stress of Disabled Athletes
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Bahar Anaforoglu, Assoc Prof, Ankara Yildirim Beyazıt University
Other Study IDs: AnkaraYBUfby
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Paralympic Athletes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months

SUMMARY:
It is aimed to investigate the relationship between anxiety, depression, stress and physical activities of disabled athletes prepared for the paralympic games to be held in Tokyo in 2021, 3 times in total at 2-3 months intervals, and to determine the change over time

ELIGIBILITY:
Inclusion Criteria:

* Being a physically disabled athlete
* Preparation for the Paralympic Games
* Volunteering to participate in the study

Exclusion Criteria:

* Serious psychiatric illness
* Regular use of sedatives or neuropsychiatric drugs
* presence of active alcohol or drug addiction
* Presence of a systemic or neurological problem that develops independent of disability pathology.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: disabled athletes who prepared the Paralympic Games
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | 8 months
  This inventory consists of two subscales(state and trait), each consisting of 20 questions. The state anxiety scale determines how the individual feels at a particular moment and under certain conditions, while the trait anxiety scale determines how the individual feels independent of the situation and conditions he or she is in.
The Center for Epidemiological Studies Depression Scale (CES-D) | 8 months
  The CES-Depression Scale is a short self-report scale developed by the American National Institute of Mental Health to be used in scientific studies to evaluate the depressive symptoms of the general population. The scale has 20 items and asks questions about feelings and thoughts about the past week.
Fatigue Severity Scale | 8 months
  It is used to determine the fatigue status of the participants. The scale consists of 9 items and evaluates the last week.
International Physical Activity Questionnaire short form | 8 months
  The questionnaire, consisting of seven questions, provides information about sitting, walking, moderately activities, and time spent on vigorous activities. The total score is calculated by adding walking, moderate-intensive, vigorous activity, and the duration (minutes) and frequency (days) of these activities
Perceived Stress Scale (PSS-14) | 8 months
  Consisting of 14 items, the PSS is designed to measure how stressful certain situations in a person's life are perceived.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt Univercity, Ankara, Turkey (Türkiye)